CLINICAL TRIAL: NCT03152448
Title: Two-Part Prospective Study to Measure Impact of Prolaris® Testing Added to Treatment Decision Following Biopsy in Newly Diagnosed Prostate Cancer Patients to Measure Prediction of Progression/Recurrence in Men Treated at VAMC
Brief Title: Prospective Prolaris Value and Efficacy
Acronym: P-PROVE
Status: Terminated | Type: Observational
Why Stopped: Myriad has sufficient data to do an analysis on the primary objective, durability, and has made the decision not to continue collecting data for the other study objectives.
Sponsor: Myriad Genetic Laboratories, Inc. (Industry)
Collaborators: VA Salt Lake City Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: URO-005
Record Dates: First submitted 2016-02-19; First posted 2017-05-15 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
Keywords: Prolaris; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Genes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Formalin-fixed paraffin-embedded (FFPE) tissue from blocks or slides of prostatic adenocarcinoma biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early Stage Prostate Cancer: Recently diagnosed treatment-naïve patients with early stage localized prostate cancer
  Interventions: Behavioral: Prolaris

INTERVENTIONS:
Behavioral: Prolaris — Series of three questionnaires to capture treatment decisions based upon standard clinical-pathological information with the addition of Prolaris genomic testing result
  Other Names: RNA expression signature based on a set of cell cycle progression (CCP) genes

SUMMARY:
This is a prospective study to measure the impact on first-line therapy of genomic testing of biopsy tissue from recently diagnosed treatment-naïve patients with early stage localized prostate cancer.

DETAILED DESCRIPTION:
This is a prospective study to measure the impact on first-line therapy of genomic testing of biopsy tissue from recently diagnosed treatment-naïve patients with early stage localized prostate cancer. Multiple individual VAMC sites will participate in PART 1 of the study. During PART 1 of the study, a three-part questionnaire will be completed to evaluate the PRE-Prolaris test treatment plan, the POST-Prolaris test treatment plan, and the ACTUAL treatment option. Using PRE-Prolaris Test Questionnaire #1 the physician will record the recommendation for first-line therapy based on standard clinical-pathological parameters (PSA, Gleason score, clinical stage and percent positive cores). The likelihood of recommending a non-interventional therapy approach will also be recorded using a 10-point ordinal scale. A sample of the biopsy tissue will then be tested using the Prolaris® genomic test and a relative cancer aggressiveness score will be shared with the physician. After reviewing and considering the results of the genomic testing and after patient consultation, the physician will complete POST-Prolaris Questionnaire #2 documenting the planned treatment ( interventional treatment or non-interventional). Approximately 6 months from the date of the test results, ACTUAL Treatment Questionnaire #3 will be completed to document the actual treatment administered.

PART 2 of this study is a prospective evaluation of the prognostic utility of Prolaris® testing of prostate biopsy samples obtained from men who participate in PART 1of the study and who undergo radical prostatectomy or radiation therapy or who are managed with WW or AS. The central VAMC site will be responsible for PART 2; individual VAMC sites will not participate in this part of the study. Patients will be followed using medical record review every 6 months for objective progression (BCR, radiographic or radionuclide evidence of metastases or disease specific mortality) through 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed (<= 6 months), untreated patients with histologically proven adenocarcinoma of the prostate
* Final treatment decision has not been made (that is all treatment options are feasible and none have been ruled out due to comorbidities at study entry)
* Clinically localized (no evidence on clinical or imaging studies of advanced disease)
* No hormonal therapy for treatment of prostate cancer including LHRH agonist or antagonist, anti-androgen, estrogens or exogenous androgens when applicable (use of 5-alpha reductase inhibitors is acceptable)
* Sufficient amount of tissue remains from biopsy to perform genomic testing
* Life expectance of a minimum of 10 years
* Men who completed PART 1 and were treated with radical prostatectomy (including robotic, laparoscopic, open retropubic or perineal) or receive radiation therapy or were placed on AS or WW.

Exclusion Criteria:

* Men with clinical node positive or metastatic disease
* Men with a known baseline total serum testosterone level of <100 ng/dL prior to radiation or hormone therapy (men with unknown baseline testosterone levels will not be excluded)
* Men who previously received pelvic radiotherapy for another malignancy
* Non adenocarcinoma prostate cancer histologies

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed, clinically localized treatment naïve prostate cancer patients in the US clinical setting
Sampling Method: Non-Probability Sample
Enrollment: 1511 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Impact of Prolaris on the magnitude of change between Pre-Prolaris treatment selection and the actual implemented treatment | 6 months
  Comparison of percentage change from the Pre-Prolaris test treatment option (based on standard clinical pathological parameters) versus the actual treatment option implemented following results of Prolaris
Prolaris prediction of biochemical or objective recurrence | 5 years
  Biochemical recurrence (defined as PSA >0.2 ng/ml or by Phoenix definition) or objective recurrences of disease by 5 years following definitive therapy with curative intent in men treatment with radical prostatectomy or radiation therapy

OTHER OUTCOMES:
Prolaris prediction of who benefits from the addition of hormone therapy to contemporary radiation therapy | 5 years
  either biochemical or objective recurrences of disease following definitive therapy with curative intent in men treated with radiation who did or did not receive adjuvant ADT
Comparison of prognostic utility of prospective Prolaris testing of prostate biopsy samples to other clinical pathological parameters with respect to disease progression | 5 years
  either biochemical or objective recurrences of disease following definitive therapy with curative intent in men treated with radical prostatectomy or radiation
Association of Prolaris score with progression to active intervention when initially managed with AS or WW | 5 years
  Progression to interventional therapy in men initially managed with AS or WW
Prognostic utility of Prolaris testing compared to other clinical pathological parameters with respect to disease progression in men who were Gleason score <7 on initial biopsy | 5 years
  biochemical or objective recurrence of disease in men who were Gleason score <7
Impact of Prolaris on magnitude of change between pre-Prolaris treatment selection and the post-Prolaris treatment plan following consultation with the patient | 3 months
  comparison of percentage change from the pre-Prolaris treatment option versus the post-Prolaris treatment plan
Impact of Prolaris on magnitude of change between physician likelihood of recommending non-interventional therapy and the likelihood following the genomic test results | 3 months
  mean change in the physician's likelihood of recommending watchful waiting or active surveillance post-genomic testing compared to pre-genomic testing

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - VA San Diego Healthcare System, San Diego, California
  - VA Connecticut Healthcare System, West Haven, Connecticut
  - James A. Haley Veterans' Hospital, Tampa, Florida
  - Kansas City VAMC, Kansas City, Kansas
  - Southeast Louisiana Veterans Healtchare System, New Orleans, Louisiana
  - Minneapolis VA Healthcare System, Minneapolis, Minnesota
  - VA St. Louis Healthcare System, St Louis, Missouri
  - James J. Peters VA, The Bronx, New York
  - Oklahoma City Veteran's Hospital, Oklahoma City, Oklahoma
  - Ralph H. Johnson VAMC, Charleston, South Carolina
  - Michael E. DeBakey VAMC, Houston, Texas
  - Salt Lake City VA Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Results of Prolaris testing to be shared with provider and patient per commercial process; study results to be presented in a pier reviewed publication in aggregate form only (no individual participant data to be shared through publications or abstracts)